CLINICAL TRIAL: NCT00875498
Title: Intermittent Theta Burst Stimulation (iTBS) for the Treatment of Negative Symptoms in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Principal Investigator, Dr. E. Poulet, PUPH, Hôpital le Vinatier
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-A00558-47
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
Keywords: iTBS; Negative Symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active iTBS (Active Comparator): iTBS active intensity = 80%MT during 6 minutes. 20 sessions, 2 per day
  Interventions: Procedure: active iTBS
- sham iTBS (Placebo Comparator): iTBS placebo (placebo coil)with same parameters than active
  Interventions: Procedure: sham iTBS

INTERVENTIONS:
Procedure: active iTBS — Intermittent Theta Burst Stimulation (iTBS) over Left dorsolateral prefrontal cortex.
  80% MT, 20 sessions of 6 minutes, 2 per day
  Other Names: TMS; rTMS; TBS; iTBS
  Arms: active iTBS
Procedure: sham iTBS — iTBS placebo (placebo coil)
  Other Names: placebo TMS; placebo rTMS
  Arms: sham iTBS

SUMMARY:
The purpose of this study is to determine whether the iTBS is an effective treatment of the negative symptoms of schizophrenia.

DETAILED DESCRIPTION:
This study will evaluate whether the intermittent Theta Burst Stimulation (iTBS), a new high frequency TMS protocol is efficient in the treatment of the Negative Symptoms of schizophrenia.

Neuroimaging studies demonstrate that hypoactivity in the left dorsolateral prefrontal cortex (LDLPFC) was associated with negative symptoms.

The investigators hypothesize that iTBS applied to LDLPFC will improve negative symptoms and will improve activity of the LDLPFC measured with Magnetic Resonance Spectroscopy (MRS).

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia according to DSM-IV
* Negative symptoms for at least 6 weeks
* Medication resistance according to Kane et al., 1988
* Age between 18 and 50 years old
* Informed consent

Exclusion Criteria:

* Contraindication to TMS
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2008-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Scale for the Assessment of Negative Symptoms (SANS) | before, after 2 weeks of treatment, and 3 times follow-up (1, 3 and 6 months)

SECONDARY OUTCOMES:
Neurochemical impact of treatment measured by 1H-MRS, DTI and resting MRI | 3 times, before treatment, immediatly after treatment and a last evaluation 3 months after

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Poulet, MD, PhD, Principal Investigator — Hopital Le Vinatier; JEROME BRUNELIN, PhD, Study Director — Hopital le Vinatier
Locations (1):
- Hopital Le vinatier, Bron, France